CLINICAL TRIAL: NCT04330898
Title: Spanish Registry of Patients With Implantable Cardiac Devices That Require a Diagnostic Imaging Test With Nuclear Magnetic Resonance
Brief Title: Patients With Implantable Cardiac Devices Requiring a Nuclear Magnetic Resonance
Acronym: RESONANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trialance SCCL (Industry)
Responsible Party: Sponsor
Other Study IDs: RMN01
Record Dates: First submitted 2019-12-09; First posted 2020-04-02 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Implantable Cardiac Device. Patients With a NMR Indication
Keywords: Peacemaker; implantable cardioverter-defibrillator; Nuclear Magnetic Resonance
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Biotronik peacemakers, implantable cardioverter-defibrillators and cardiac resynchronizers — Any of these Biotronik cardiac stimulation devices with the Home Monitoring function activated for the remote control of patients

SUMMARY:
The general objective of this registry is to study the number of patients carrying an implantable cardiac device that have an indication for an imaging diagnosis based on nuclear magnetic resonance. Is wanted to know the cause of the indication of the diagnostic test based on MRI.

DETAILED DESCRIPTION:
MRI is currently infra indicated in patients with cardiac stimulation devices and for this reason, the request for this imaging technique in these patients is complicated and, often, the MRI-based test is replaced by a CT scan that may not be so beneficial for the diagnosis.

Current data indicate that, with cardiological control and maintaining basic safety precautions, MRI could be performed in patients with peacemakers and Implantable Cardioverter Defibrillators (ICD) that require it for clinical reasons, although it should be noted that currently, due to lack of data published, the absolute safety of an MRI in these patients and the protocol used in each case cannot be guaranteed.

This registry proposal is to have data of all patients implanted with Biotronik cardiac stimulation devices and evaluate how many of them have an indication for an MRI-based diagnostic test, how many of them are already undergoing this diagnostic test, how many are given an tomography as an alternative to avoid subjecting patients to an MRI

ELIGIBILITY:
Inclusion Criteria:

* Patients carrying a cardiac stimulation device
* Patients able to understand the nature of the procedure
* Patients who give informed consent

Exclusion Criteria:

* Epicardial cables
* Abandoned cables
* Non-BIOTRONIK cables
* Age <18 years
* Pregnant and breastfeeding
* Subjects with irreversible brain damage caused by a pre-existing brain disease
* Heart transplant 6 months prior to recruitment or expected within the next 3 months
* Cardiac surgery 3 months prior to recruitment or planned for the next 3 months
* Life expectancy less than 12 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with an accepted indication of an implantable cardiac device, including pacemakers, defibrillators and cardiac resynchronizers
Sampling Method: Probability Sample
Enrollment: 1248 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with implantable cardiac devices that require a diagnostic test based on MRI | 1 year
  statistical analysis of the variable

SECONDARY OUTCOMES:
Primary indication for MRI | 1 year
  statistical analysis of the variable
Reasons for not used MRI | 1 year
  statistical analysis of the variable
Percentage of patients with a non-MRI-based test diagnosis, although they had an indication for an MRI-based diagnostic test because of their disease | 1 year
  statistical analysis of the variable
Cost effectiveness of the he MRI Autodetect function | 1 year
  statistical analysis of the variable
Analysis of the differences in the workflow | 1 year
  statistical analysis of the variable

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Alzueta, MD, PhD, Principal Investigator — Hospital Virgen de la Victoria; Francisco Ruiz Mateas, MD, PhD, Principal Investigator — Hospital Costa del Sol
Locations (20):
- Spain (20):
  - Hospital San Pedro de Alcantara, Cáceres, Madrid
  - Hospital de Poniente, El Ejido, Madrid
  - Hospital Arquitecto Marcide, Ferrol, Madrid
  - Hospital de Galdakano, Galdakao, Madrid
  - Hospital de Orense, Orense, Madrid
  - Hospital General de Asturias, Oviedo, Madrid
  - Hospital Virgen del Puerto, Plasencia, Madrid
  - Hospital de Puerto Real, Puerto Real, Madrid
  - Hospital Parc Taul'i, Sabadell, Madrid
  - Hospital Marques de Valdecilla, Santander, Madrid
  - Hospital Rio Hortega, Valladolid, Madrid
  - Hospital Universitatis de Araba, Vitoria, Madrid
  - Hospital General de Alicante, Alicante
  - Hospital San Juan de Alicante, Alicante
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marcu CB, Beek AM, van Rossum AC. Clinical applications of cardiovascular magnetic resonance imaging. CMAJ. 2006 Oct 10;175(8):911-7. doi: 10.1503/cmaj.060566. PMID 17030942
- [Background] Durack DT, Lukes AS, Bright DK. New criteria for diagnosis of infective endocarditis: utilization of specific echocardiographic findings. Duke Endocarditis Service. Am J Med. 1994 Mar;96(3):200-9. doi: 10.1016/0002-9343(94)90143-0. PMID 8154507
- [Background] Kanal E, Borgstede JP, Barkovich AJ, Bell C, Bradley WG, Etheridge S, Felmlee JP, Froelich JW, Hayden J, Kaminski EM, Lester JW Jr, Scoumis EA, Zaremba LA, Zinninger MD; American College of Radiology. American College of Radiology White Paper on MR Safety: 2004 update and revisions. AJR Am J Roentgenol. 2004 May;182(5):1111-4. doi: 10.2214/ajr.182.5.1821111. No abstract available. PMID 15100103
- [Result] Gold MR, Sommer T, Schwitter J, Al Fagih A, Albert T, Merkely B, Peterson M, Ciuffo A, Lee S, Landborg L, Cerkvenik J, Kanal E; Evera MRI Study Investigators. Full-Body MRI in Patients With an Implantable Cardioverter-Defibrillator: Primary Results of a Randomized Study. J Am Coll Cardiol. 2015 Jun 23;65(24):2581-2588. doi: 10.1016/j.jacc.2015.04.047. Epub 2015 May 14. PMID 25982014